CLINICAL TRIAL: NCT01434238
Title: Evaluation of an Infant Feeding Support Strategy for HIV-exposed Infants 6-12 Months Old in Urban Haiti
Brief Title: Evaluation of an Infant Feeding Intervention for HIV-exposed Haitian Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic (Other); Weill Medical College of Cornell University (Other); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB 0907000316
Record Dates: First submitted 2011-09-09; First posted 2011-09-14 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Lack of; Care, Infant (Child), Malnutrition
Keywords: infant feeding; HIV; growth; anemia
MeSH Terms: conditions — Malnutrition; Anemia | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention participant (Experimental)
  Interventions: Other: Counseling and nutrition supplement

INTERVENTIONS:
Other: Counseling and nutrition supplement — 24-week intervention that includes a) a daily ration of fortified lipid-based nutrient supplement and b) nutrition counseling delivered through biweekly group and individualized sessions. Dietary supplement is a locally- produced lipid-based nutrient spread (Meds and Foods for Kid, Cap Haitian, Haiti) that in a 65g daily ration provides 345 kcal energy and single allowance of key micronutrients for the 6-12 month age group.

SUMMARY:
The purpose of this quasi-experimental study is to evaluate the effectiveness of an infant feeding intervention in improving growth and anemia outcomes among HIV-exposed infants 6-12 months of age.

DETAILED DESCRIPTION:
The need for better nutrition during infancy to improve growth and child survival outcomes is well recognized and is especially acute in the context of maternal human immunodeficiency virus (HIV) infection. WHO Guidelines on Infant Feeding and HIV call for support of HIV-infected caregivers during infant feeding transitions across the first year of life. However, there are few published examples of programmatic approaches that effectively integrate PMTCT and infant feeding support at the service delivery level.

The objectives of this study are to develop and test an infant feeding support intervention among non-breastfed HIV-exposed infants age 6-12 months enrolled in the Prevention of Mother-to-Child Transmission of HIV program at the GHESKIO centres, an HIV and TB treatment clinic in urban Port-au-Prince, Haiti. The investigators hypothesize that growth and anemia outcomes will be better in the intervention cohort compared to historical controls. The investigators also hypothesize that the infant feeding support intervention will be feasible and acceptable to mothers and clinical staff.

To accomplish these objectives, the investigators will enroll 82 HIV-exposed infants age 5.5-6.5 months recruited from the GHESKIO pediatric clinic in a 24-week intervention that includes a) a daily ration of fortified lipid-based nutrient supplement and b) nutrition counseling delivered through biweekly group and individualized sessions. Data on growth, supplement use, infant feeding knowledge and practices will be collected every 4 weeks during the intervention period. Hemoglobin and dietary intake will be assessed at baseline, mid-point and end of intervention. Intervention children will be seen 6-months post intervention to assess growth and anemia outcomes. Growth and anemia outcomes in the intervention group will be compared to medical record data from same-age HIV-exposed children seen at GHESKIO in the previous year.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed maternal HIV-infection
* Age 5.5-6.5 months at intervention start
* Weight-for-length z-score > -3 SD (WHO 2006 reference)

Exclusion Criteria:

* Confirmed or suspected allergy to peanuts
* Participation in a concurrent clinical trial at GHESKIO

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in prevalence of growth faltering during the intervention | end of intervention (approximately 12 months of age)
  Change in weight-for-age, length-for-age and weight-for-length <-2 SD based on WHO 2006 Growth Standard
Change in prevalence of growth faltering post-intervention | Six-months post-intervention (approximately 18 months of age)
  Change in weight-for-age, length-for-age and weight-for-length <-2 SD based on WHO 2006 Growth Standard

SECONDARY OUTCOMES:
Change in prevalence of anemia during intervention | end of intervention (approximately 12 months of age)
  Prevalence of anemia (Hb < 10.5 g/dl)
Dietary intake | end of intervention (approximately 12 months of age)
  dietary nutrient intakes assessed through 24-hour dietary recall

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Heidkamp, PhD, Principal Investigator — Cornell University
Locations (1):
- GHESKIO Centres, Port-au-Prince, Quest, Haiti

REFERENCES:
- [Derived] Heidkamp RA, Stoltzfus RJ, Fitzgerald DW, Pape JW. Growth in late infancy among HIV-exposed children in urban Haiti is associated with participation in a clinic-based infant feeding support intervention. J Nutr. 2012 Apr;142(4):774-80. doi: 10.3945/jn.111.155275. Epub 2012 Feb 29. PMID 22378328